CLINICAL TRIAL: NCT01594658
Title: Prospective Random Study for Handling Venous Ulcer With Conservative Treatment (Dressings Alone) and Foam Sclerotherapy Versus Conservative Treatment
Brief Title: Venous Ulcer Treatment With Foam Versus Conservative Treatment
Acronym: VUTEF
Status: Completed | Type: Observational
Sponsor: Hospital Occidente de Kennedy (Other)
Collaborators: Universidad El Bosque, Bogotá (Other)
Responsible Party: Principal Investigator, ernesto nieves, medical doctor, Hospital Occidente de Kennedy
Other Study IDs: VUT-3F
Record Dates: First submitted 2011-07-18; First posted 2012-05-09 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Venous Ulcer
Keywords: Ultrasound-guided foam sclerotherapy; chronic venous ulcers
MeSH Terms: conditions — Varicose Ulcer | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Foam sclerotherapy: This arm corresponds to ultrasound-guided foam sclerotherapy of superficial venous reflux plus conservative management
  Interventions: Procedure: Foam sclerotherapy
- Conservative: This arm only has medical standard handling (healings performed by the nurse group)
  Interventions: Procedure: conservative

INTERVENTIONS:
Procedure: Foam sclerotherapy — Foam application of 1% (Sklerol®, ICV Pharma, Bogota-Colombia), Reg INVIMA: 2002M-0001016, guided by ecography of insufficient superficial veins, doses from 10-40 cc of foam until obtaining endoluminal occlusion of the vein. The patient will rest for 8 minutes and then the leg will be covered with elastic bandage.
  Other Names: (Sklerol®, ICV Pharma, Bogota-Col),Reg INVIMA: 2002M-0001016
  Groups: Foam sclerotherapy
Procedure: conservative — This arm only has medical standard handling (healings performed by the nurse group)
  Other Names: This arm only has medical standard handling
  Groups: Conservative

SUMMARY:
The venous ulcer due to venous insufficiency causes an important morbility to those people suffering from this condition. Most of therapies available under the obligatory health plan (POS, acronym in spanish) to date cover the cleaning of the ulcerous lesion and its medical handling using saline solutions, topical antibiotics and elastic dressings, implying an important intake from health resources due to its chronicity and the delay in ulcers healing, which usually takes periods ranging from 6 months to several years. therapeutical alternatives, which can guarantee optimal, fast and persistent in time healings, should be identified.

The aim of this study is to determine the percentage of healing of active venous ulcers (using a clinical, etiological, anatomic and physiopathologic classification (CEAP), C6) following ultrasound-guided foam sclerotherapy of superficial venous reflux in patients with chronic venous ulceration after six months from the intervention, compared with conservative medical handling. The investigators expect that the ultrasound-guided foam sclerotherapy of superficial venous reflux will diminish the time of ulcer healing compared with standard handling.

DETAILED DESCRIPTION:
to determine healing rates following ultrasound-guided foam sclerotherapy (UGFS) of superficial venous reflux (SVR) in patients with open (clinical,etiologic, anatomic and pathophysiologic (CEAP) classification, C6) chronic venous ulceration ( CVU) in a randomised clinical trial of foam sclerotherapy for patients with venous ulcer

ELIGIBILITY:
Inclusion Criteria:

* Presence of Venous Ulcer confirmed by CEAP C6
* Chronic venous ulcer present for at least 4 weeks
* Ankle-arm index greater or equal to 0.8 mmHg

Exclusion Criteria:

* Severe hepatic, cardiac or pulmonary disease
* Deep venous thrombosis
* Active participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with C6 by CEAP Clasification
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Venous Ulcer Treatment with Foam Versus Conservative Treatment | 6 months
  Number of participants with healing of venous ulcer after six months from the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Ramirez, MD, Study Director — Hospital Occidente de Kennedy
Locations (1):
- Hospital Occidente de Kennedy, Bogota, Cundinamarca, Colombia

REFERENCES:
- [Background] Pang KH, Bate GR, Darvall KA, Adam DJ, Bradbury AW. Healing and recurrence rates following ultrasound-guided foam sclerotherapy of superficial venous reflux in patients with chronic venous ulceration. Eur J Vasc Endovasc Surg. 2010 Dec;40(6):790-5. doi: 10.1016/j.ejvs.2010.08.011. Epub 2010 Sep 27. PMID 20875753
- [Background] Darvall KA, Bate GR, Adam DJ, Silverman SH, Bradbury AW. Ultrasound-guided foam sclerotherapy for the treatment of chronic venous ulceration: a preliminary study. Eur J Vasc Endovasc Surg. 2009 Dec;38(6):764-9. doi: 10.1016/j.ejvs.2009.05.027. Epub 2009 Jul 18. PMID 19616975